CLINICAL TRIAL: NCT02823171
Title: A Phase 1, Open-Label, Single-Dose, Randomized, 2-Period Crossover Study to Assess the Bioequivalence of Two Pacritinib Drug Product Formulations (Phase 3 Clinical Trial [P3CT] Formulation [Reference] and Final Market Image [FMI] Formulation [Test]) Following Oral Administration in Healthy Subjects
Brief Title: To Assess the Bioequivalence of Two Pacritinib Drug Product Formulations and FMI Formulation Following Oral Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PAC108
Record Dates: First submitted 2016-05-03; First posted 2016-07-06 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Bioequivalence Study; Healthy subjects

ARMS (2):
- Sequence I (Experimental): Sequence I: treatment A/B
  Interventions: Drug: Treatment A: 400 mg Pacritinib P3CT; Drug: Treatment B: 400 mg of pacritinib FMI
- Sequence II (Experimental): Sequence II: treatment B/A
  Interventions: Drug: Treatment A: 400 mg Pacritinib P3CT; Drug: Treatment B: 400 mg of pacritinib FMI

INTERVENTIONS:
Drug: Treatment A: 400 mg Pacritinib P3CT — 400-mg oral dose of pacritinib P3CT (reference) formulation capsules
  Other Names: PAC400mg P3CT
Drug: Treatment B: 400 mg of pacritinib FMI — 400-mg oral dose of pacritinib FMI (test) formulation capsules
  Other Names: PAC400mg FMI

SUMMARY:
A Phase 1, Open-Label, Single-Dose, Randomized, 2-Period Crossover Study to Assess the Bioequivalence of Two Pacritinib Drug Product Formulations (Phase 3 Clinical Trial [P3CT] Formulation [Reference] and Final Market Image [FMI] Formulation [Test]) Following Oral Administration in Healthy Subjects

DETAILED DESCRIPTION:
This study will be a Phase 1, open-label, single-dose, randomized, 2-period, 2-treatment sequence crossover study to determine the bioequivalence of pacritinib following administration of 400-mg doses of P3CT (Reference) and FMI (Test) formulations and to characterize the PK of pacritinib.

Each subject will receive 2 treatments (a 400-mg oral dose of four 100-mg pacritinib P3CT [reference] formulation capsules and a 400-mg oral dose of four 100-mg pacritinib FMI [test] formulation capsules) in a 2-period crossover design. Each treatment will be administered as monotherapy during 1 of 2 treatment periods. A 9-day washout will separate the 2 administrations of study medication. Subjects will remain confined to the Clinical Research Unit (CRU) throughout the study for safety observation and PK blood sample collection

ELIGIBILITY:
Inclusion Criteria:

1. males or females, aged 18 to 55 years, inclusive, who are not tobacco users;
2. with BMI in the range of 18.0 to 32.0 kg/m2, inclusive;
3. in good health, determined by no clinically significant findings from medical history, physical examination, and vital signs as determined by the Investigator, in consultation with the sponsor;
4. normal 12-lead ECG, or ECG findings (including RR, PR, and QT intervals; QT interval corrected using Fridericia's formula [QTcF]; QRS duration; and ventricular heart rate) deemed not clinically significant by the Investigator, in consultation with the Sponsor;
5. clinical laboratory evaluations (including clinical chemistry panel [fasted at least 10 hours], CBC, and UA) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator, in consultation with the Sponsor; laboratory values may be confirmed by repeat;
6. negative test for selected drugs of abuse (including alcohol) at Screening and at Check-in (Day -1 of Period 1);
7. negative hepatitis panel (including HBsAg and anti-HCV) and negative HIV antibody screens;
8. females of childbearing potential must not be pregnant or lactating, and must agree to use 1 of the following forms of contraception from the time of signing the informed consent or 10 days prior to Check-in (Day -1) of Period 1 until 30 days after the final dose administration: non-hormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; intravaginal system (eg, NuvaRing®); diaphragm with spermicide; cervical cap with spermicide; male sexual partner who agrees to use a male condom with spermicide; sterile sexual partner; or abstinence. Oral, implantable, transdermal, or injectable hormonal contraceptives may not be used from the time of signing the informed consent or 10 days prior to Check-in (Day -1) of Period 1 until 14 days after the final dose administration. For all females, the pregnancy test result must be negative at Screening and Check-in (Day -1) of Period 1. Females not of childbearing potential must be postmenopausal for at least 1 year or surgically sterile (eg, tubal ligation, hysterectomy) for at least 90 days;
9. males will be surgically sterile (ie, vasectomy, documented in the medical record by a physician) or agree to use, from Check-in (Day -1) of Period 1 until 90 days following Study Completion/ET, 1 of the following approved methods of contraception: male condom with spermicide; sterile sexual partner; or use by female sexual partner of an IUD with spermicide, a female condom with spermicide, a contraceptive sponge with spermicide, an intravaginal system, a diaphragm with spermicide, a cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives. Subjects must agree to refrain from sperm donation from Check-in (Day -1) of Period 1 until 90 days following Study Completion/ET;
10. able to comprehend and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

1. prior ingestion of pacritinib;
2. history or clinical manifestation of clinically significant cardiovascular, pulmonary, hepatic (eg, hepatitis), renal, hematologic, gastrointestinal (eg, celiac disease, peptic ulcer, gastroesophageal reflux, inflammatory bowel disease), metabolic, allergic, dermatological, neurological, or psychiatric disorder (as determined by the Investigator; appendectomy and cholecystectomy are not considered to be clinically significant events);
3. significant abnormalities in liver function tests (alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase >1.5 × upper limit of normal [ULN]; gamma-glutamyl transferase >2 × ULN; or total bilirubin >1.3 × ULN) or kidney function tests (serum creatinine > ULN) that are considered clinically significant by the Investigator; laboratory values may be confirmed by repeat;
4. history of malignancy, except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps;
5. history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator in consultation with the Sponsor;
6. history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy, cholecystectomy, and hernia repair will be allowed;
7. history of Gilbert's Syndrome;
8. history or presence of ECG QTcF >450 msec, factors that increase risk for QTc interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome);
9. history of alcoholism or drug addiction within 1 year prior to Check-in (Day -1) of Period 1;
10. use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1) of Period 1 and during the entire study;
11. consumption of alcohol- or caffeine-containing foods and beverages for 72 hours prior to Screening and during the entire study;
12. consumption of grapefruit-containing foods and beverages or other CYP3A4 inhibitors or inducers for 72 hours prior to Screening and during the entire study;
13. subjects will refrain from strenuous exercise from 48 hours prior to Check-in (Day -1) of Period 1 and during the period of confinement at the CRU and will otherwise maintain their normal level of physical activity throughout the entire study (ie, will not begin a new exercise program nor participate in any unusually strenuous physical exertion);
14. participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days prior to Check-in (Day -1) of Period 1, whichever is longer, and during the entire study;
15. female subjects who are unable to refrain from the use of oral, implantable, injectable, or transdermal hormonal contraceptives within 10 days prior to Check-in (Day -1) of Period 1 or from the time of signing the informed consent until 14 days after the final dose administration;
16. use of any prescription medications and/or products within 14 days prior to Check-in (Day -1) of Period 1 and during the entire study, unless deemed acceptable by the Investigator, in consultation with the Sponsor;
17. use of any over-the-counter, non-prescription medications (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in (Day -1) of Period 1 and during the entire study, unless deemed acceptable by the Investigator, in consultation with the Sponsor;
18. poor peripheral venous access;
19. donation of blood from 30 days prior to Screening through Study Completion/ET, inclusive, or plasma from 2 weeks prior to Screening through Study Completion/ET, inclusive;
20. receipt of blood products within 2 months prior to Check-in (Day -1) of Period 1;
21. any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The apparent total body clearance (CL/F) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib were assessed following 400 mg single-dose administration of Clinical trial material or final market image formulations of pacritinib capsule in healthy subjects
The maximum plasma concentration (Cmax). | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib were assessed following 400 mg single-dose administration of Clinical trial material or final market image formulations of pacritinib capsule in healthy subjects
The area under the plasma concentration-time curve from time zero to time of the last measured concentration above the limit of quantification (AUC0-t). | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib were assessed following 400 mg single-dose administration of Clinical trial material or final market image formulations of pacritinib capsule in healthy subjects
The area under the plasma concentration-time curve from zero to infinity (AUC0-∞). | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib were assessed following 400 mg single-dose administration of Clinical trial material or final market image formulations of pacritinib capsule in healthy subjects
The time to reach maximum plasma concentration (tmax). | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib were assessed following 400 mg single-dose administration of Clinical trial material or final market image formulations of pacritinib capsule in healthy subjects
The apparent volume of distribution (Vd) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib were assessed following 400 mg single-dose administration of Clinical trial material or final market image formulations of pacritinib capsule in healthy subjects

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Day 1 to Day 17
  Safety and tolerability of pacritinib 400 mg

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Whitehurst, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit Inc., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes